CLINICAL TRIAL: NCT01959295
Title: Phase III Study of ASP2151 in Herpes Simplex Patients - A Double-blind, Placebo-controlled Study -
Brief Title: Phase III Study of ASP2151 in Herpes Simplex Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Maruho Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M522101-J11
Record Dates: First submitted 2013-09-26; First posted 2013-10-10 (Estimated); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Herpes Simplex
MeSH Terms: conditions — Herpes Simplex | interventions — ASP2151

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ASP2151 (Experimental)
  Interventions: Drug: ASP2151
- ASP2151 placebo (Placebo Comparator)
  Interventions: Drug: ASP2151 placebo

INTERVENTIONS:
Drug: ASP2151 — 200 mg once daily
  Arms: ASP2151
Drug: ASP2151 placebo — once daily
  Arms: ASP2151 placebo

SUMMARY:
To evaluate the efficacy and safety of ASP2151 in patients with herpes simplex.

DETAILED DESCRIPTION:
A double-blind, randomized, placebo-controlled, parallel-group study will be conducted to evaluate the efficacy and safety of ASP2151 in patients with herpes simplex (labial/facial herpes or recurrent genital herpes). The efficacy will be evaluated for the primary endpoint defined as, "the proportion of subjects achieving lesion healing by Day 8 of study treatment" to demonstrate the superiority of ASP2151 to placebo. The safety will be evaluated based on adverse events, laboratory tests, vital signs, and ECGs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a rash associated with moderate or severe herpes simplex, for which oral antiviral medication is indicated

   * Labial/facial herpes: Patients with at least 10 papulae or vesicles/pustules
   * Recurrent genital herpes: Patients with at least 5 papulae or vesicles/pustules on the genital organs or in the genital and circumanal region
2. Patients who can start receiving the study drug within 48 hours after onset of rash
3. Age: 20 years or older, but younger than 80 years

Exclusion Criteria:

1. Patients who are not expected to have an adequate response to oral antiviral medication
2. An extreme decline in immune function
3. Presence of serious complications
4. Patients found to meet any of the following conditions based on laboratory tests performed within 14 days before informed consent:

   * AST or ALT ≥ 2.5 x upper limit of normal
   * Platelet count < lower limit of normal
   * Serum creatinine ≥ 1.5 mg/dL
   * Creatinine clearance < 30 mL/min
5. Current or previous history of malignant tumor within 5 years before informed consent
6. Diagnosis of autoimmune disease
7. Evidence of bone marrow suppression

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2013-08; Primary Completion 2015-04 (Actual); Study Completion 2015-04-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (3):
  - Sapporo, Hokkaido
  - Yokohama, Kanagawa
  - Nakano-ku, Tokyo

RESULTS

PARTICIPANT FLOW:
Groups:
- ASP2151 Placebo: ASP2151 placebo once daily
Period: Overall Study
Arm/Group | ASP2151 | ASP2151 Placebo
Started | 311 | 157
Completed | 278 | 140
Not Completed | 33 | 17
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 0 | 2
Not completed — Physician Decision | 2 | 3
Not completed — Protocol Violation | 16 | 5
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Clinical laboratory value is ineligible on day 1 | 10 | 6

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS). The FAS was defined as patients who were diagnosed with labial/facial herpes or recurrent genital herpes at the time of case registration, subsequently received the study drug at least once, and had any efficacy variable measured, except for those found not to have herpes simplex after study drug administration.
Groups:
- ASP2151: 200mg once daily
- Total: Total of all reporting groups
Arm/Group | ASP2151 | ASP2151 Placebo | Total
Number analyzed (Participants) | 307 | 154 | 461
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 287 | 147 | 434
  >=65 years | 20 | 7 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (12.9) | 40.5 (13.5) | 40.4 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 219 | 107 | 326
  Male | 88 | 47 | 135
Region of Enrollment [Number; unit: participants]
  Japan | 307 | 154 | 461
Disease type [Count of Participants; unit: Participants]
  Labial/facial herpes | 264 | 133 | 397
  Recurrent genital herpes | 43 | 21 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Healing by Day 8
Description: The percentage of participants achieving lesion healing by Day 8 of study treatment
Time Frame: 8days
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Arm/Group | ASP2151 | ASP2151 Placebo
Number analyzed (Participants) | 307 | 154
Percentage of Participants | 66.4 | 69.5
Statistical Analysis 1: Comparison: ASP2151 vs ASP2151 Placebo; The superiority of ASP2151 200mg to ASP2151 placebo was assessed by Mantel-Haenszel method, adjusted by disease type (labial/facial herpes and recurrent genital herpes); Test type: Superiority; p = 0.5086, Mantel Haenszel

2. Secondary Outcome: Time to Healing
Description: The criteria for determining healing are as follows:
  1. A condition where all erythematous and papular lesions, vesicular and pustular lesions, and erosive and ulcerative lesions have been resolved, and either the complete resolution of crusts or the complete epithelialization beneath any remaining crusts has been achieved.
  2. In participants where no crust has formed, a condition characterized by the epithelialization of erosions/ulcers formation in mucosal lesions and potentially other affected areas.
  3. In participants where no vesicles or pustules have formed, a condition characterized by the complete resolution of all erythematous and papular lesions
Time Frame: 29days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | ASP2151 | ASP2151 Placebo
Number analyzed (Participants) | 307 | 154
day | 8 [6 to 9] | 8 [6 to 9]

3. Secondary Outcome: Time to Complete Crusting
Description: The criteria for complete crust formation are outlined as follows:
  1. A condition where all erythematous and papular lesions, vesicular and pustular lesions, and erosive and ulcerative lesions have been resolved, and all rashes are crusted (epithelialization beneath is not required).
  2. In participants where no crust has formed, a condition characterized by the epithelialization of erosions/ulcers formation in mucosal lesions and potentially other affected areas.
  3. In participants where no vesicles or pustules have formed, a condition characterized by the complete resolution of all erythematous and papular lesions.
Time Frame: 29days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | ASP2151 | ASP2151 Placebo
Number analyzed (Participants) | 307 | 154
day | 6 [5 to 8] | 6 [5 to 8]

4. Secondary Outcome: Time to Virus Disappearance
Description: The day of viral disappearance is the first day on which the results of viral isolation continuously show 'HSV negative' until the final implementation day. The negative means that the results of the isolation and culture are negative, or the isolation and culture has not been performed due to complete crusting or healing of the lesion site.
Time Frame: 29days
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: day
Arm/Group | ASP2151 | ASP2151 Placebo
Number analyzed (Participants) | 307 | 154
day | 4 [3 to 6] | 5 [4 to 6]

ADVERSE EVENTS:
Time Frame: 29 days
Description: The safety analysis population consists of 466 participants (309 in the ASP group;157 in the placebo group), excluding two participants who were randomized but never received the investigational drug.
  The two excluded participants were discontinued from the study before receiving the investigational drug, and therefore, they were not monitored or assessed for adverse events.
Arm/Group | ASP2151 | ASP2151 Placebo
All-Cause Mortality (participants affected / at risk) | 128/309 | 59/157
Serious Adverse Events (participants affected / at risk) | 0/309 | 0/157
Other Adverse Events (participants affected / at risk) | 69/309 | 29/157
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ASP2151 (N=309) | ASP2151 Placebo (N=157)
Genital herpes (Infections and infestations) | 11 | 3
Nasopharyngitis (Infections and infestations) | 15 | 5
Oral herpes (Infections and infestations) | 13 | 8
Beta-N-acetyl-D-glucosaminidase increased (Investigations) | 9 | 2
Electrocardiogram QT prolonged (Investigations) | 3 | 4
Fibrin degradation products increased (Investigations) | 13 | 4
Alpha 1 microglobulin increased (Investigations) | 23 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes